CLINICAL TRIAL: NCT00791895
Title: NovoLog® Mix 70/30 (Biphasic Insulin Aspart 70/30) Titrate-To-Target: An Observational Study of the Efficacy of NovoLog® Mix 70/30 in Patients With Type 2 Diabetes Mellitus Not Achieving Glycemic Targets on OADs With / Without Once Daily Basal Insulin Therapy
Brief Title: Efficacy of Biphasic Insulin Aspart 30 in Type 2 Diabetics Failing on OADs
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BIASP-2174
Record Dates: First submitted 2008-11-13; First posted 2008-11-17 (Estimated); Last update posted 2017-02-24 (Actual); Status verified 2017-02

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — insulin aspart, insulin aspart protamine drug combination 30:70; Insulin Aspart

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Experimental)
  Interventions: Drug: biphasic insulin aspart 30

INTERVENTIONS:
Drug: biphasic insulin aspart 30 — Treat-to-target dose titration scheme
  Other Names: BIASP; NovoLog® Mix 70/30; NovoMix®

SUMMARY:
This trial is conducted in the United States of America (USA). The aim of this trial is to investigate the effectiveness of biphasic insulin aspart 30 in type 2 diabetics not achieving blood sugar levels when treated with oral anti-diabetics drugs (OADs) with or without basal insulin therapy.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes mellitus for at least 12 months
* HbA1c: 7.5-10.0%
* An antidiabetic regimen that has been stable for at least 3 months
* Able and willing to perform SMBG testing as per protocol

Exclusion Criteria:

* Use of any insulin preparations other than NPH or glargine within the past 6 months
* Pregnancy, breastfeeding, intention to become pregnant within the next 12 months, or judged to be using inadequate contraceptive measures (adequate contraceptive measures includes: sterilization, intrauterine devices, oral contraceptives, or consistent use of barrier methods)
* Known or suspected allergy to trial product or agents related to trial product

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2003-06-26 (Actual); Primary Completion 2004-10-31 (Actual); Study Completion 2004-11-29 (Actual)

PRIMARY OUTCOMES:
Percentage of subjects achieving HbA1c below 6.5% | after 16, 32 and 48 weeks, respectively

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (14):
- United States (14):
  - Novo Nordisk Investigational Site, Phoenix, Arizona
  - Novo Nordisk Investigational Site, La Jolla, California
  - Novo Nordisk Investigational Site, DeLand, Florida
  - Novo Nordisk Investigational Site, Wichita, Kansas
  - Novo Nordisk Investigational Site, Omaha, Nebraska
  - Novo Nordisk Investigational Site, Albany, New York
  - Novo Nordisk Investigational Site, Cleveland, Ohio
  - Novo Nordisk Investigational Site, Medford, Oregon
  - Novo Nordisk Investigational Site, Memphis, Tennessee
  - Novo Nordisk Investigational Site, Dallas, Texas
  - Novo Nordisk Investigational Site, Houston, Texas
  - Novo Nordisk Investigational Site, Ogden, Utah
  - Novo Nordisk Investigational Site, Renton, Washington
  - Novo Nordisk Investigational Site, Milwaukee, Wisconsin

REFERENCES:
- [Result] Garber AJ, Wahlen J, Wahl T, Bressler P, Braceras R, Allen E, Jain R. Attainment of glycaemic goals in type 2 diabetes with once-, twice-, or thrice-daily dosing with biphasic insulin aspart 70/30 (The 1-2-3 study). Diabetes Obes Metab. 2006 Jan;8(1):58-66. doi: 10.1111/j.1463-1326.2005.00563.x. PMID 16367883
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com